CLINICAL TRIAL: NCT04027413
Title: A Double-Blind, Randomised, Placebo-Controlled Trial of Protein Supplementation to Enhance Exercise Capacity in Chronic Obstructive Pulmonary Disease
Brief Title: Protein Supplementation to Enhance Exercise Capacity in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Nutricia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 18/LO/1842
Record Dates: First submitted 2019-06-27; First posted 2019-07-22 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: COPD
Keywords: Pulmonary Rehabilitation; Nutrtional supplements
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants will be randomised using a web-based service called 'sealed envelope' and stratified BMI less and equal or more than 20 kg/m2 to control group or interventional group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant in both groups will received either the supplement or the placebo/ control products. Both products will be labelled the same way.
  Investigator: someone not from the research team will run the randomisation and deliver the products to participants.
  Outcome Assessor: will not be involved in the randomisation and will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo/ Control (Placebo Comparator): participants in this group will receive carbohydrate product which does not include protein at all
  Interventions: Dietary Supplement: preOp
- Intervention group (Experimental): Participants in this group will receive high protein product
  Interventions: Dietary Supplement: fortisip compact protein

INTERVENTIONS:
Dietary Supplement: fortisip compact protein — (24% protein; 41% carbohydrate; 35% fat)
  Arms: Intervention group
Dietary Supplement: preOp — (100% carbohydrate).
  Arms: Placebo/ Control

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common smoking-related lung disease.

Pulmonary Rehabilitation (PR) is a six-week supervised group exercise and education class. PR is an effective intervention in COPD to reduce symptoms, improve exercise performance and prevent exacerbation. Exercise intolerance/limitation is one of the commonest issues with COPD patients and this may be compounded by reduced muscle mass and malnutrition. COPD patients lose body weight and skeletal muscle mass which leads to muscle weakness and dysfunction, thus impacting functional ability and quality of life. Muscle weakness is caused by a prolonged sedentary lifestyle and voluntary immobilization. Importantly, being under-weight is associated with an increased risk of mortality in COPD.

Nutritional supplementation have been used to overcome malnutrition in COPD patients. It has been shown that nutritional support integrated with exercise training can improve exercise activity, decreased the risk of mortality, and improve muscle strength in undernourished COPD patients. However, uptake of nutritional supplementation during pulmonary rehabilitation, where the potential benefit may be greatest, has been limited by the absence of rigorous evidence-based studies supporting use.

Investigators want to investigate the effect of a nutritional supplement during a PR program on exercise capacity in COPD patients. Investigators will collect demographic data, distribute questionnaires, measure exercise performance, and some additional measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed COPD (post-bronchodilator forced vital capacity in one second: forced vital capacity ratio <0.7)
2. >10 smoking pack year history.
3. Enrolling on a pulmonary rehabilitation programme.
4. Age of 18 and above.

Exclusion Criteria:

1. Patients with any physical or mental health disorders preventing compliance with trial protocol.
2. Unable to communicate in English
3. Malabsorption syndrome
4. Unable to perform the Incremental Shuttle Walk Test
5. Patients already using other types of oral dietary supplement, under the care of a dietitian.
6. Galactosaemia (contraindication)
7. Known cow's milk protein allergy or lactose intolerance
8. BMI >30kg/m2 without recent weight loss of >5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 12 weeks
  The difference in change of exercise capacity before and and after pulmonary rehabilitation between intervention and control groups measured by Incremental Shuttle Walk Test.

SECONDARY OUTCOMES:
Peripheral muscle strength | 12 weeks
  The difference in change of peripheral muscle strength Before and and after pulmonary rehabilitation between intervention and control groups measured by Hand Dynamometer.
Rectus femoris muscle cross-sectional | 12 weeks
  The difference in change of Rectus femoris muscle cross-sectional area before and and after pulmonary rehabilitation between intervention and control groups measured by portable ultrasound.
Body composition | 12 weeks
  The difference in change of body composition fat mass (FM) before and and after pulmonary rehabilitation between intervention and control groups measured by a device called Bodystat.
Physical activity | 14 days
  The difference in change of physical activity before and and after pulmonary rehabilitation between intervention and control groups measured by step-counter (YAMAX SW200).
Health-related quality of life | 12 weeks
  The difference in change of health-related quality before and after pulmonary rehabilitation between intervention and control groups measured by Hospital Anxiety and Depression Scale. consists of seven items for anxiety and seven items for depression, each item has a score from 0-3.This means that a person can score between 0 and 21 for either abnormal, respectively. 0-7 = Normal, 8-10 = Borderline abnormal and 11-21 = Abnormal
Body circumferences | 12 weeks
  The difference in change of waist circumference before and and after pulmonary rehabilitation between intervention and control groups measured by a tape.
Body composition | 12 weeks
  The difference in change of body composition fat free mass (FFM) before and and after pulmonary rehabilitation between intervention and control groups measured by a device called Bodystat.
Body composition | 12 weeks
  The difference in change of body composition fat free mass index (FFMI) before and and after pulmonary rehabilitation between intervention and control groups measured by a device called Bodystat.
Body circumferences | 12 weeks
  The difference in change of hip circumference before and and after pulmonary rehabilitation between intervention and control groups measured by a tape.
Body circumferences | 12 weeks
  The difference in change of mid-thigh circumference before and and after pulmonary rehabilitation between intervention and control groups measured by a tape.
Health-related quality of life | 12 weeks
  The difference in change of health-related quality before and after pulmonary rehabilitation between intervention and control groups measured by the COPD Assessment Test Questionnaire.
Health-related quality of life | 12 weeks
  The difference in change of health-related quality before and after pulmonary rehabilitation between intervention and control groups measured by St. George's Respiratory Questionnaire.
intervention compliance | 6 weeks
  participants intervention compliance will be assessed by sheet
Food intake | 12 weeks
  Food intake for 3 consecutive days before, during, and after PR by food diary
Lower limb function | 12 weeks
  The difference in change of lower limb function before and after pulmonary rehabilitation between intervention and control groups measured Sit to Stand - Five Test.
Malnutrition risk | 12 weeks
  The difference in change of Malnourished risk before and after pulmonary rehabilitation between intervention and control groups measured Malnutrition Universal Screening Tool .
Disability associated with breathlessness | 12 weeks
  The difference in change of Disability associated with breathlessness before and after pulmonary rehabilitation between intervention and control groups measured by Medical Research Council breathlessness scale .
Body weight | 12 weeks
  The difference in change of body weight before and after pulmonary rehabilitation between intervention and control groups measured by digital scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Central and North West London Foundation Trust, London, United Kingdom